CLINICAL TRIAL: NCT02926339
Title: Teens Against Tobacco Use: A Tobacco Prevention Curriculum and Advocacy Initiative
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: El Paso Independent School District (Unknown); Paso del Norte Health Foundation (Other)
Responsible Party: Principal Investigator, Louis D. Brown, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HSC-SPH-16-0534
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Tobacco Smoking Behavior
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teens Against Tobacco Use presentation (Experimental): Students in the intervention group will receive anti-tobacco presentations from Teens Against Tobacco Use Members
  Interventions: Behavioral: Teens Against Tobacco Use presentation
- Control (No Intervention): Students in this group will receive a control presentation from their physical education teachers on a topic unrelated to tobacco.

INTERVENTIONS:
Behavioral: Teens Against Tobacco Use presentation — Students receive a series of 3 anti-tobacco presentations delivered by older peers
  Arms: Teens Against Tobacco Use presentation

SUMMARY:
This study evaluates the efficacy of Teens Against Tobacco Use anti-tobacco presentations on tobacco use susceptibility in 6th through 8th grade. Students will be randomly assigned to either receive 3 anti-tobacco presentations or 3 presentations on a different topic, unrelated to tobacco.

DETAILED DESCRIPTION:
The investigators will collaborate with Austin High School, Wiggs Middle School, and Guillen Middle School of the El Paso Independent School District to implement smoke free youth coalitions as an after school activity. The coalitions will follow the Teens Against Tobacco Use (TATU) model developed by the American Lung Association, the American Cancer Society, and the American Heart Association. Participating youth will be trained to develop and deliver anti-tobacco presentations to younger students. Each school will have a separate youth coalition operating under the guidance of an adult coordinator. High school youth will present to middle school classes, whereas middle school youth will present to 4th and 5th graders.

To evaluate the efficacy of the TATU program, we will randomly assign students in physical education classes to receive TATU presentations or a control condition. Confidential surveys about tobacco will be administered at the beginning and end of the school year. Analyses will compare intervention and control students on smoking susceptibility, perceptions of harm from tobacco use, tobacco industry perceptions, and social norms on tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Students from participating schools
* 6th to 8th grade students
* Classes must be willing to receive presentations in the fall and spring semesters.

Exclusion Criteria:

* Students from non-participating schools
* Students not able to read English or Spanish

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 639 (Actual)
Dates: Start 2016-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Tobacco Susceptibility assessed by Likert scale questions drawn primarily from the global youth tobacco survey | Change from Baseline Tobacco Susceptibility at 7 months
  Tobacco susceptibility captures the likelihood of using tobacco in the future. It will be assessed by likert scale questions drawn primarily from the global youth tobacco survey. It will be analyzed as a continuous variable that will be standardized, so outcomes will represent standard deviation unit differences in tobacco susceptibility.

CONTACTS AND LOCATIONS:
Overall Officials: Louis D Brown, PH.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, School of Public Health, El Paso Regional Campus, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided